CLINICAL TRIAL: NCT01967368
Title: Safety and Efficacy of Intradermal Trivalent Influenza Vaccination in Institutionalized Older Adults
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Chan Tuen Ching, Resident Specialist, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UW 12339
Record Dates: First submitted 2013-10-16; First posted 2013-10-22 (Estimated); Last update posted 2013-10-22 (Estimated); Status verified 2013-10

CONDITIONS: Influenza, Human
Keywords: Influenza vaccine; intradermal; intramuscular; efficacy; safety
MeSH Terms: conditions — Influenza, Human | interventions — vaxigrip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intanza (Experimental): intradermal injection (15ug hemagglutinin 2013/2014 trivalent influenza vaccine) delivered with the Intanza, single dose injection
  Interventions: Drug: Intanza
- Vaxigrip (Active Comparator): intramuscular injection (15ug hemagglutinin 2013/2014 trivalent influenza vaccine) delivered with the Vaxigrip, single dose injection
  Interventions: Drug: Vaxigrip

INTERVENTIONS:
Drug: Intanza — Principal Investigator would be responsible for injecting the intradermal vaccine in a sterile technique.
  Other Names: Intanza, intradermal trivalent influenza vaccine
  Arms: Intanza
Drug: Vaxigrip — Principal Investigator would be responsible for injecting the intrmuscular vaccine in a sterile technique.
  Other Names: Vaxigrip, intramuscular trivalent influenza vaccine
  Arms: Vaxigrip

SUMMARY:
Influenza is associated with significant morbidity and mortality. Institutionalized older adults (age>65) is the group associated with highest risk of complications. Influenza vaccines are the cornerstone of influenza prevention but one systematic review has found that there is no statistically significant difference against laboratory confirmed influenza. A major reason is immune senescence in older adults which result in weaker response towards vaccines when compared with young adults. Intradermal administration of vaccine has been suggested to improve immune response due to the abundance of immunostimulatory cells, such as dendritic cells in the dermis. Intradermal administration of influenza vaccine has been shown to have comparable or superior efficacy compared with intramuscular administration in the >60-year old population and the rates of adverse events post-vaccination were also comparable between them. The immunogenicity of intradermal administration has also been shown to be better in immunocompromised patients, including community dwelling older adults. In addition, intradermal vaccination has good acceptability and safety profile in different countries, so it has been licensed in Hong Kong and worldwide. However, there is little study regarding the efficacy of intradermal vaccination of influenza in institutionalized older adults, investigators therefore would like to perform a prospective, randomized study to compare the safety and immunogenicity between conventional full dose intramuscular immunization and full dose intradermal immunization of the trivalent influenza vaccine in institutionalized older adults.

The hypothesis is that full dose intradermal trivalent influenza vaccination is as effective as full-dose standard intramuscular injection in terms of seroconversion and seroprotection rate in institutionalized older adults. Finding of this study will be important in the vaccination of institutionalized older adults and immunocompromised patients as intradermal vaccine may induce a better immune response against influenza infection.

DETAILED DESCRIPTION:
This is a prospective, randomized, parallel-group single centre trial in the Queen Mary Hospital and Fung Yiu King Hospital. Investigators aim to recruit 100 subjects who would be qualified for the Hospital Authority (HA)/ Centre for Health Protection (CHP) Mass Vaccination Program for Trivalent influenza vaccine (TIV). These patients include Institutionalized older adult patients at the age of 65 or above.

After informed consent (allow patient one week to consider) subjects will be randomly assigned into 2 groups to receive the following vaccines: Group 1: the full-dose (1 dose) standard TIV (15ug hemagglutinin TIV) delivered intramuscularly using a conventional needle, Group 2: a full-dose (1 dose) intradermal injection (15ug hemagglutinin TIV) delivered with the Intanza 15 at day 0. All TIV vaccines used in this study will be either of Vaxigrip® (Group 1) or Intanza® Intradermal (Group 2), Sanofi-Pasteur and provided by the Hospital Authority or the University of Hong Kong. Baseline HI to the TIV will be measured at day 0.

Patients fulfilling the inclusion criteria will be screened from the Community Geriatric Assessment Team (CGAT) of Fung Yiu King Hospital by the investigators. Before commencing, patients would be allowed to have one week to consider joining the study. Meanwhile, investigators would also take 5ml of serum from the participant to test for the baseline TIV antibody. Principal Investigator is experienced in administering intramuscular injections and he would be responsible for refilling the low-dose intradermal injection in a sterile technique. The microneedle device used in this study comprises an array of three 0.6 mm microneedles, made up of silicon crystal, and bonded to the tip of a plastic adapter, which can be mounted on any standard syringe. During injection, the microneedle device was lightly pushed against the shoulder so that the microneedles penetrated the outmost layer of skin. The entire vaccine dose will then be injected causing a blanched bleb to appear. Intramuscular injection of conventional full-dose vaccine is given in the usual way with the prefilled syringe. Principal Investigator will be responsible for subject bleeding, serum separation, storing in doublet copies, freezing and archiving, according to HKU protocols.

MN and HI analysis (see below) shall be conducted by the HKU Laboratory according to the following protocols:

Microneutralization antibody assay (MN) NT will be performed inside a type II Biosafety Cabinet in a Biosafety Containment level III facility. NT will be performed in 96-well microtiter plates seeded with MDCK cells. Two fold serial dilutions of paired serum (pre- and post-vaccination) will be tested in duplicates against 100 TCID50 of the following 3 viruses: A/California/7/2009 (H1N1)pdm09-like virus; an A/Victoria/361/2011 (H3N2)-like virus; and a B/Wisconsin/1/2010-like virus in the presence of L-1-tosylamide-2-phenylethyl chloromethyl ketone (TPCK)-treated trypsin (TPCK-trypsin; Sigma). A corresponding set of cell controls with sera but without virus inoculation will be used as controls. The cells will be scored for the inhibition of the cytopathic effect (CPE) at 72~96 hours. The titer of neutralization antibody is defined as the maximum dilution of serum at which the percentage of CPE is less than or equal to 50%.

HI assay Serum samples will be tested for Hemagglutination inhibition (HI) antibody against the following: A/California/7/2009 (H1N1)pdm09-like virus; an A/Victoria/361/2011 (H3N2)-like virus; and a B/Wisconsin/1/2010-like virus using reference antigens (WHO influenza reagent kit provided by the World Health Organization influenza Collaborating Centre, CDC, Atlanta, Georgia, USA. HAI antibody assays will be performed by standard microtiter techniques after removal of non-specific inhibitors in serum with receptor destroying enzyme (RDE) (1:3), incubation overnight at 37 degree C followed by heat-inactivation at 56 degree C for 30 minutes. All serum samples from each subject will be tested for each of the test antigens. Serial two-fold dilutions of RDE-treated serum from 1:10 will be titrated against 4 hemagglutinin units of reference antigens using 0.25% turkey erythrocytes. A doublet backup of each serum sample would be prepared and frozen in two separately located freezers at -20ºC for potential future analysis and/or validation.

Outcome measures:

Primary outcome:

a. Change from baseline (day 0 of vaccination )in neutralization antibody titre against influenza at day 21 and day 180 of vaccination

Secondary outcomes:

a. Adverse effects at day 0-7

ELIGIBILITY:
Inclusion Criteria:

* Institutionalized older adult patients at the age of 65 or above

Exclusion Criteria:

* Clinically significant immune-related diseases and significant recent co-morbidities

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-05 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in neutralization antibody titre against influenza | day 0 (baseline), day 21 and day 180 of vaccination
  Neutralization antibody titre against the 3 influenza viruses are tested 3 times at day 0, day 21 and day 180 of vaccination for comparison. The titer of neutralization antibody is defined as the maximum dilution of serum at which the percentage of cytopathic effect is less than or equal to 50%.

SECONDARY OUTCOMES:
Adverse effects | day 0 and day 7 of vaccination
  Adverse effects due to vaccination from day 0 to day 7 will be recorded. Adverse effects boardly divided into local and systemic. Local adverse effect include swelling, erythema, pruritis, pain. Systemic adverse effect include fever, malaise, myalgia

CONTACTS AND LOCATIONS:
Overall Officials: Tuen Ching Chan, MBBS, Principal Investigator — The University of Hong Kong, Department of Medicine, Queen Mary Hospital
Locations (1):
- Queen Mary Hospital and Fung Yiu King Hospital, Hong Kong West Cluster, Hospital Authority, Hong Kong, China

REFERENCES:
- [Derived] Chan TC, Hung IF, Chan KH, Li CP, Li PT, Luk JK, Chu LW, Chan FH. Immunogenicity and safety of intradermal trivalent influenza vaccination in nursing home older adults: a randomized controlled trial. J Am Med Dir Assoc. 2014 Aug;15(8):607.e5-12. doi: 10.1016/j.jamda.2014.05.002. Epub 2014 Jun 21. PMID 24957950